CLINICAL TRIAL: NCT03668366
Title: S-1 Combined With IMRT Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoshen Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-S1-02
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; IMRT; S-1
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-1 arm (Experimental): The patients in the S-1 arm will receive IMRT (66-70.4Gy to GTV, 57-60.8Gy to CTV1, 54-56Gy to CTV2, given in 30-32 fractions). During the IMRT course, S-1 will be administered orally according to body surface area (BSA<1.25m2, 30mg; BSA: 1.25-1.5m2, 40mg; BSA>1.5m2, 50mg) twice per day for 30-32 days. The dose modifications of S-1 will not be permitted during concurrent chemotherapy unless progression of the disease, toxicities of grade 4 or patient's refusal.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — The patients will receive IMRT combined with S-1 concurrent chemoradiotherapy. The specific treatment description is included in arm description.

SUMMARY:
This study is a prospective phase II trial which is designed to evaluate the efficacy and safety of IMRT combined with S-1 CCRT for locally advanced NPC. Eligibility criteria include histologically confirmed locally advanced NPC according to the American Joint Committee on Cancer (AJCC) Staging System (the eighth edition); Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; at least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1; normal complete blood count, normal hepatic function and normal renal function. Prior induction chemotherapy with platinum was allowed.

Exclusion criteria include previous radiotherapy, a history of any other type of malignancy; pregnancy or lactation; allergy to S-1; obvious dysfunction of liver, renal, cardiac or lung function; uncontrolled infection; systemic metastasis or distant metastasis; patients with severe gastrointestinal diseases, and patients with mental disorders affecting patient participation in trial judgement.

The full-set pretreatment evaluation will be performed to every patient.All patients in this study will receive intensity-modulated radiation therapy (IMRT). During the IMRT course, S-1 will be administered orally according to body surface area.The dose modifications of S-1 will not be permitted during concurrent chemotherapy unless progression of the disease, toxicities of grade 4 or patient's refusal.

The primary endpoints of this study is adverse events (AE) rate and progression-free survival (PFS).

DETAILED DESCRIPTION:
This study is a prospective phase II trial which is designed to evaluate the efficacy and safety of IMRT combined with S-1 CCRT for locally advanced NPC. Eligibility criteria include histologically confirmed locally advanced NPC according to the American Joint Committee on Cancer (AJCC) Staging System (the eighth edition); Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; at least one measurable lesion based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1; normal complete blood count (white blood cell counts ≥4×1012/L, hemoglobin level ≥100g/L and platelet counts ≥100×1012/L), normal hepatic function (total bilirubin level ≤1.5 mg/dl, alanine aminotransferase and aspartate aminotransferase levels ≤1.5 times the upper limit of normal) and normal renal function (creatinine ≤ 1.5 times the upper limit of normal). Prior induction chemotherapy with platinum was allowed.

Exclusion criteria include previous radiotherapy, a history of any other type of malignancy; pregnancy or lactation; allergy to S-1; obvious dysfunction of liver, renal, cardiac or lung function; uncontrolled infection; systemic metastasis or distant metastasis; patients with severe gastrointestinal diseases, and patients with mental disorders affecting patient participation in trial judgement.

The full-set pretreatment evaluation will be performed to every patient.All patients in this study will receive intensity-modulated radiation therapy (IMRT). During the IMRT course, S-1 will be administered orally according to body surface area (BSA<1.25m2, 30mg; BSA: 1.25-1.5m2, 40mg; BSA>1.5m2, 50mg).The dose modifications of S-1 will not be permitted during concurrent chemotherapy unless progression of the disease, toxicities of grade 4 or patient's refusal.

Adverse events (AEs) will be evaluated every week during CCRT based on the evaluation criteria of adverse reactions of CTCAE V4.0. Tumor response is assessed at the end of CCRT according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1. Radiation-related acute and late toxicities are graded according to the Radiation Therapy Oncology Group (RTOG). Late toxicities are evaluated beyond three months from the end of radiotherapy.

After the completion of CCRT, all patients will be followed up every 3 months during the first years, every 6 months for the following 2-5 years, and annually thereafter. Local recurrence is confirmed by nasopharynx MRI or histological biopsy. Regional recurrence is confirmed by fine needle aspiration or surgical biopsy. Distant metastases is detected by imaging examinations including PET-CT, bone Emission Computed Tomography (ECT), CT, MRI or confirmed by histological confirmation of biopsy.

The primary endpoints of this study is adverse events (AE) rate and progression-free survival (PFS). PFS is calculated from the date of enrollment to the date of disease progression or the date of death for any cause.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced NPC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Normal complete blood count
* Normal hepatic function
* Normal renal function (creatinine ≤ 1.5 times the upper limit of normal).

Exclusion Criteria:

* Previous radiotherapy
* A history of any other type of malignancy
* Pregnancy or lactation
* Allergy to S-1
* Obvious disfunction of liver, renal, cardiac or lung function
* Uncontrolled infection
* Systemic metastasis or distant metastasis
* Patients with severe gastrointestinal diseases
* Patients with mental disorders affecting patient participation in trial judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
PFS | 3-year PFS （2018-2021）
  PFS is calculated from the date of the enrollment to the date of disease progression or the date of death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshen Wang, MD,Ph.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China